CLINICAL TRIAL: NCT01305538
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Cross-over Study of the Efficacy and Safety of BMS-954561 in Patients With Post-herpetic Neuralgia (PHN)
Brief Title: Crossover Post-herpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CN169-002; 2010-023041-30 (EudraCT Number)
Record Dates: First submitted 2011-02-14; First posted 2011-02-28 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Post-Herpetic Neuralgia (PHN)
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 BMS-954561 40mg or 80mg (Other): Arm description: BMS-954561 40mg or 80mg three times daily (TID) to Placebo OR Placebo to 40mg or 80mg TID.
  Arm type: Active to Placebo or Placebo to Active (cross-over)
  Interventions: Drug: BMS-954561; Drug: Placebo
- Arm 2 BMS-954561 150mg or 300mg (Other): Arm description: BMS-954561 150mg or 300mg TID to Placebo OR Placebo to 150mg or 300mg TID
  Arm type: Active to Placebo or Placebo to Active(cross-over)
  Interventions: Drug: BMS-954561; Drug: Placebo

INTERVENTIONS:
Drug: BMS-954561
  Arms: Arm 1 BMS-954561 40mg or 80mg
Drug: BMS-954561
  Arms: Arm 2 BMS-954561 150mg or 300mg
Drug: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of study drug (BMS-954561) as compared to placebo in the treatment of patients with post-herpetic neuralgia (PHN).

DETAILED DESCRIPTION:
Allocation: Randomized Stratified

Interventional model: Cross-over Placebo Controlled

ELIGIBILITY:
Inclusion Criteria:

* Patient with Post-Herpetic Neuralgia (PHN) as defined as pain present for more than 6 months after the onset of a herpes zoster skin rash affecting the trigeminal, cervical, thoracic, lumbar, or sacral regions.
* Based on patient diary information collected during the Baseline week (day -7 to randomization Day 1), patient has completed at least 5 diary entries and has an average weekly pain rating of at least 4 on the 11-point pain rating scale.
* The patient is able to satisfactorily complete, in the Investigator's judgment, the Cognitive Battery.
* Male or female, 18-85 years of age.

Exclusion Criteria:

* Other severe pain that may potentially confound pain assessment.
* History of complete lack of response to pregabalin (at least 300 mg qd for 4 weeks) or gabapentin (at least 1800 mg qd for 4 weeks).
* Hemoglobin A1c > 9%
* Hemoglobin ≤ 9 g/dL.
* Active herpes zoster or known viral infection.
* Previous neurolytic or neurosurgical therapy for PHN.
* Estimated glomerular filtration rate (eGFR) according to the re-expressed abbreviated (four-variable) Modification of Diet in Renal Disease (MDRD) Study equation ≤ 40ml/min/1.73m2.
* Patients who have been on a stable dose of anticonvulsant,anticholinergic, antiviral medications, nicotine replacements, or any other smoking cessation medications for <4 weeks prior to randomization. Patients who are on stable doses for => 4 weeks prior to randomization are allowed, however, there should be no adjustments to the dose of these medications during study.
* Patients currently on more than one drug for treatment of neuropathic pain (low dose opioids, antidepressants, or anticonvulsants). Patients are allowed to participate if on a stable dose for at least 4 weeks prior to randomization (Day1) and should remain stable during course of study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the average pain score for BMS-954561 vs. placebo. | up to 10 weeks

SECONDARY OUTCOMES:
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Screening/Baseline Phase: Baseline
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 1
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 2
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 3
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 4
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 5
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 6
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 7
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 8
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 9
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Weeks 10
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Weeks 2
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Weeks 4
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Weeks 8
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Weeks 12
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Weeks 16
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Weeks 20
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 1
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 2
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 3
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 4
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 5
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 6
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 7
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 8
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 9
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Weeks 10
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Weeks 2
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Weeks 4
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Weeks 8
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Weeks 12
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Weeks 16
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Weeks 20
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Screening/Baseline Phase: Baseline
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 1
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 2
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 3
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 4
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 5
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 6
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 7
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 8
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 9
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Weeks 10
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Weeks 2
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Weeks 4
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Weeks 8
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Weeks 12
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Weeks 16
Evaluate the tolerability and safety of BMS-954561 in patients with post-herpetic neuralgia as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Weeks 20

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (19):
  - Arizona Research Center, Phoenix, Arizona
  - Torrance Clinical Research, Lomita, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Brain Matters Research, Delray Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, Llc, Orlando, Florida
  - Comprehensive Clinical Development, Inc., St. Petersburg, Florida
  - Drug Studies America, Marietta, Georgia
  - Commonwealth Biomedical Research, Llc, Madisonville, Kentucky
  - Analgesic Solutions, Natick, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - The Center For Pharmaceutical Research. Pc, Kansas City, Missouri
  - Medex Healthcare Research, Inc, St Louis, Missouri
  - Finger Lakes Clinical Research, Rochester, New York
  - Wake Research Associates, Llc, Raleigh, North Carolina
  - Pmg Research Of Winston-Salem, Winston-Salem, North Carolina
  - Radiant Research, Inc., Akron, Ohio
  - Cor Clinical Research, Oklahoma City, Oklahoma
  - Futuresearch Trials Of Neurology, Austin, Texas
- France (4):
  - Local Institution, Bordeaux
  - Local Institution, Boulogne-Billancourt
  - Local Institution, Nice
  - Local Institution, Saint-Priest-en-Jarez

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx